CLINICAL TRIAL: NCT04222933
Title: Effect of Motorized Cryotherapy on Early Effusion, Swelling, and Pain After Anterior Cruciate Ligament Reconstruction: a Randomized Controlled Trial
Brief Title: Effect of Motorized Cryotherapy on Early Effusion, Swelling, and Pain After Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanyang University Seoul Hospital (Other)
Responsible Party: Principal Investigator, JIN KYU LEE, professor, Hanyang University Seoul Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Hanyang university cryo
Record Dates: First submitted 2020-01-05; First posted 2020-01-10 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Cryotherapy Effect

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motorized cryotherapy (Experimental): Application of motorized cryotherapy after ACL reconstruction for 6 postoperative days
  Interventions: Device: Motorized cryotherapy
- Classical cryotherapy (Active Comparator): Application of ice bags for 6 postoperative days
  Interventions: Device: Classical cryotherapy

INTERVENTIONS:
Device: Motorized cryotherapy — application of motorized cryotherapy after ACL reconstruction
  Arms: Motorized cryotherapy
Device: Classical cryotherapy — application of an ice bag
  Arms: Classical cryotherapy

SUMMARY:
To test the efficacy of motorized cryotherapy on early effusion, and pain after ACL reconstruction

DETAILED DESCRIPTION:
To test the efficacy of motorized cryotherapy on early effusion, and pain after ACL reconstruction compared to classical ice bagging

ELIGIBILITY:
Inclusion Criteria:

* Acute ACL ruptured patient

Exclusion Criteria:

* Combined meniscal injury requiring surgery
* Combined ligament injury requiring surgery
* Combined chondral injury requiring surgery
* Previous surgery history on corresponding knee
* Allergic to cold

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Pain after surgery | postoperative day 4
  VAS pain scale (0 to 10 points, higher the worse pain)

SECONDARY OUTCOMES:
Effusion after surgery | baseline, postoperative day 4, 7, 14, 6 weeks
  Effusion by thigh circumference (cm), MRI measurement (cc)

CONTACTS AND LOCATIONS:
Overall Officials: JIN KYU LEE, PHD, Principal Investigator — Hanyang University
Locations (1):
- Department of Orthopaedic Surgery, Hanyang University, College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No